CLINICAL TRIAL: NCT03275506
Title: A Randomized, Open-label, Multicentric Phase II Trial of PEMBROLIZUMAB (Keytruda®) With Chemotherapy Versus Chemotherapy Alone (Standard of Care) as Neo Adjuvant Treatment of Ovarian Cancer Not Amenable to Front Line Debulking Surgery.
Brief Title: PEMBRO With Chemo in Neo Adj Treatment of Ovarian Cancer .
Acronym: NEOPEMBROV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OV126b
Record Dates: First submitted 2017-07-18; First posted 2017-09-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer Stage IV
Keywords: neoadjuvant; debulking surgery
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: open-label, multicentric
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab + Chemotherapy (Experimental): Arm B (n=60): 4 neo-adjuvant cycles of standard 3 weekly Pembrolizumab 200 mg then carboplatin (AUC5 or 6) and paclitaxel (175mg/m²)
  Arm B: Pembrolizumab 200 mg then carboplatin (AUC5 or 6) and paclitaxel (175mg/m²), +/- bevacizumab (15 mg/kg Q3W)
  The total number of cycles of chemotherapy will be 6 cycles from the start of the neo-adjuvant chemotherapy. Three additional cycles are allowed if required (maximum 9 cycles in total).
  The planning of administration or not of bevacizumab will be defined before the randomization and could not be modified (stratification factor).
  After chemotherapy:
  * In the Arm A & B, for patients receiving bevacizumab (as standard therapy) (15 mg/kg Q3W), this will be continue until a maximum of 15 months in total from the beginning of the adjuvant therapy.
  * In the arm B, patient will receive Pembrolizumab 200 mg until a maximum of 15 months in total from the beginning of the adjuvant therapy.
  Interventions: Drug: Pembrolizumab Injectable Product - Chemotherapy - Bevacizumab
- Chemotherapy alone (Active Comparator): Arm A (n=30): 4 neo-adjuvant cycles of standard 3 weekly carboplatin (AUC5 or 6) and paclitaxel (175mg/m²)
  Arm A: carboplatin (AUC5 or 6) and paclitaxel (175mg/m²), q3 weeks +/- bevacizumab (15 mg/kg Q3W)
  The total number of cycles of chemotherapy will be 6 cycles from the start of the neo-adjuvant chemotherapy. Three additional cycles are allowed if required (maximum 9 cycles in total).
  The planning of administration or not of bevacizumab will be defined before the randomization and could not be modified (stratification factor).
  After chemotherapy:
  - In the Arm A & B, for patients receiving bevacizumab (as standard therapy) (15 mg/kg Q3W), this will be continue until a maximum of 15 months in total from the beginning of the adjuvant therapy.
  Interventions: Drug: Chemotherapy - Bevacizumab

INTERVENTIONS:
Drug: Pembrolizumab Injectable Product - Chemotherapy - Bevacizumab — Pembrolizumab 200 mg then carboplatin (AUC5 or 6) and paclitaxel (175mg/m²), +/- bevacizumab (15 mg/kg Q3W)
  Arms: Pembrolizumab + Chemotherapy
Drug: Chemotherapy - Bevacizumab — Carboplatin (AUC5 or 6) and paclitaxel (175mg/m²), +/- bevacizumab (15 mg/kg Q3W)
  Arms: Chemotherapy alone

SUMMARY:
There are several data suggesting that pembrolizumab and bevacizumab may be synergistic. Enhanced tumor angiogenesis is commonly associated with absence of tumor-infiltrating T cells in patients. There is evidence in OC that tumor expression of VEGF is negatively correlated to the density of CD3+TILs and this phenotype is associated with early recurrence, consistent with prior studies showing a correlation of VEGF to early recurrence and short survival. Furthermore, in ascites, high levels of VEGF correlate to low numbers of NK T-like CD3+CD56+ cells

This randomized phase II study aims to evaluate the efficacy of pembrolizumab in combina-tion with the standard neo adjuvant chemotherapy followed by IDS and the safety of this strategy in patients with advanced ovarian cancer. We assume that its administration in the neo adjuvant setting combination with standard of care (4 cycles of standard chemotherapy) would improve the response rate and consequently will help to achieve optimal debulking rate at IDS.

After surgery, patients will continue to be treated with standard of care (chemotherapy for 2 to 5 cycles plus or less bevacizumab) or the same combination plus pembrolizumab (keytruda).

DETAILED DESCRIPTION:
The standard procedure for initial diagnosis recommends the realization of laparoscopy first for all suspicious advanced ovarian carcinoma. This procedure should able to confirm histo-logical diagnosis and to describe the all abdominal extension of the disease.

For advanced stages, complete primary cyto-reductive surgery followed by 6 cycles of chemotherapy based remains the standard of care as first treatment in ovarian cancer. It is part of a large surgery including total hysterectomy, bilateral salpingo-oophorectomy, omentectomy, appendectomy, lymphadenectomy and removal of all peritoneal carcinomatosis.

More recently, complete resection of all macroscopic disease at primary debulking surgery has been shown to be the single most important independent prognostic factor in advanced ovarian carcinoma , and this was confirmed for interval debulking surgery (IDS) after neo adjuvant chemotherapy in the EORTC-GCG study . These results suggest that neo-adjuvant chemotherapy followed by surgical cytoreduction is an acceptable management strategy for patients with advanced ovarian cancer and is more and more frequently used in Europe in advanced ovarian cancer patients with high burden of tumor . Due to these confirmed results, the rate of patients receiving neo adjuvant chemotherapy increased over time compared to up front surgery Hence, we hypothesize that improving the response rate to neo adjuvant chemotherapy would improve the optimal debulking rate at IDS and ultimately the survival. This change of medical practices over time opened the possibility to explore new agent in combination with chemotherapy. For patients whose extent of disease is not amenable to complete or optimal upfront debulking surgery, neo adjuvant treatment with carboplatin plus paclitaxel should be considered, followed by an interval debulking surgery. A minimum of 3 cycles of carboplatin/paclitaxel must be administered before to propose interval surgery. After interval surgery, completion of the chemotherapy with 3 or 4 more chemotherapy regimen is proposed.

For patients with macroscopic residual disease or when disease remains unresectable, combination with bevacizumab to adjuvant chemotherapy then a maintenance phase of bevacizumab alone can be proposed as a standard of care Given that facts, there is a strong rationale to introduce additional neo adjuvant therapies that would strengthen the tumor shrinkage and improve the resectability rate.

Furthermore, immune surveillance plays an important role in tumor outcome of ovarian cancer patients. Indeed, clinical data in ovarian cancer patients have demonstrated that an antitumor immune response and immune evasion mechanisms are correlated, respectively, with a better and lower survival). Thus, immunotherapies are emerging as potential strategies to enhance classical EOC treatments.

More recently, they also have demonstrated significant efficacy in aggressive cancers of other histology such as metastatic Lung Cancer , metastatic Renal Cell Cancer or metastatic Bladder Cancer .

Approximately half of OC patients display a spontaneous antitumor immune response by antibodies and oligoclonal T-cells which recognize autologous tumor-associated antigens (TAAs). OC exhibits an extreme degree of heterogeneity of TAAs with an average of 60 private nonsynonymous mutations per tumor which are rarely shared among different tumors.

Though data remains scarce, high IHC PD-L1 expression (score 2 & 3) has been detected in 68% of ovarian cancer patients (n=70) and that expression of PD-L1 had a strong prognostic value . The authors found also that the density of intraepithelial CD8+ T cells was inversely correlated to expression of PD-L1 by tumors, suggesting that the expres-sion of PD-L1 on tumor cells may inhibit invasion of tumor epithelium by CD8+ T cells.

In addition, PD-1 expression at the surface of intra-tumoral CD4+ FOXP3+ Tregs was found to show the highest levels in ovarian cancer (around 20% of the cells) compared to other tumor types, including melanoma, renal cell cancer or hepatoma . Thus targeting PD-1/PD-L1 pathway may inhibit Treg expression, one of the major component of ovarian cancer immunosuppression. Also Curiel et al showed that myeloid dendritic cells (MDCs) from ovarian cancer express PD-1 and that blockade of PD-1 enhanced MDC-mediated T-cell activation, including upregulation of IL-2 and interferon-gamma, and down regulation of IL-10, which resulted in enhanced T-cell immunity against autologous ovarian human tumors into NOD-SCID mice.

Together with the aforementioned data on immune infiltration, these data provide the rationale for a therapeutic PD-1/PD-L1 pathway blockade in ovarian cancer.

In ovarian carcinoma patients, the anti-PD1 compound nivolumab has been reported to achieve 3 objectives responses out of 13 (23%) heavily pre-treated patients. Response was prolonged over 1 year in 2 out of the 3 responders. Similarly, the anti-PD1 pembrozilumab achieved 3 confirmed responses (11.5% [(95% CI, 2.4-30.2]) in 26 patients treated in a phase IB study and 3 additional patients had a tumor reduction of at least 30%. Most common AEs were fatigue (42.3%), anemia (30.8%), and decreased appetite (30.8%). Drug-related AEs occurred in 69.2% of pts (grade ≥ 3, 1/26 pts).

The anti-PD-L1 avelumab has reported a 10.7% objective response and a 44% stabilization rate in 75 patients with ovarian cancer in relapse. In this study, con-firmed or unconfirmed responses (n=11) tend to be more frequently observed in patients with low burden of tumor, limited number of prior lines of chemotherapy and in the setting of platinum-sensitivity. Toxicity was minimal. Considering all grades, fatigue was observed in 16% of the patients, chills in 12%, nausea in 10.7%, diarrhea in 10.7%, rash in 8% and hypothyroidism in 5.3%.

Rationale for combining pembrolizumab and standard chemotherapy Kryczek et al compared the PD-1 expression level at the surface of intra-tumoral CD4+ FOXP3+ Tregs among many cancer types. Interestingly, the higher level of PD-1 expression (around 20%) was found on Tregs of ovarian cancers whereas it was much lower (<10%) in other cancer types (Colon cancer, Hepatic cancer, Melanoma, Pancreatic carcinoma, Renal cell carcinoma). PD-L1 expression has also been detected in ovarian cancer tissue analysis by Immunohistochemistry staining and its level of expression has been correlated to a bad outcome of patients (59). Together with the aforementioned data on immune infiltration, these results provide rationale for a therapeutic PD-1/PD-L1 pathway blockade in ovarian cancer. In the published trials on such compounds, addition of pembrolizumab to chemotherapy or using alone has been shown to improve the response rates with a median time to response at 8 weeks (60,61).

Rationale for combining pembrolizumab and bevacizumab There are several data suggesting that pembrolizumab and bevacizumab may be synergistic. Enhanced tumor angiogenesis is commonly associated with absence of tumor-infiltrating T cells in patients. There is evidence in OC that tumor expression of VEGF is negatively correlated to the density of CD3+TILs and this phenotype is associated with early recurrence, consistent with prior studies showing a correlation of VEGF to early recurrence and short survival. Furthermore, in ascites, high levels of VEGF correlate to low numbers of NK T-like CD3+CD56+ cells.

This randomized phase II study aims to evaluate the efficacy of pembrolizumab in combina-tion with the standard neo adjuvant chemotherapy followed by IDS and the safety of this strategy in patients with advanced ovarian cancer. We assume that its administration in the neo adjuvant setting combination with standard of care (4 cycles of standard chemotherapy) would improve the response rate and consequently will help to achieve optimal debulking rate at IDS.

After surgery, patients will continue to be treated with standard of care (chemotherapy for 2 to 5 cycles plus or less bevacizumab) or the same combination plus pembrolizumab (keytruda).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Woman ≥ 18 and ≤ 75 years old on day of signing informed consent
3. Histologically confirmed diagnosis of epithelial ovarian carcinoma or fallopian tube carcinoma or primary peri-toneal carcinoma with the exception of mucinous histology. Histology should be obtained by laparoscopy (or by laparotomy).
4. High grade serous or endometrioid (see appendix 1 bis)
5. Advanced FIGO stage IIIC to IV patient not able to receive primary debulking surgery for which neo adjuvant chemotherapy with carboplatin and paclitaxel is recommended (primary debulking surgery has been denied after an evaluation through laparoscopy or laparotomy). Patients with extra abdominal metastasis (FIGO 2014 Stage IV) can be included in case of completely resectable metastasis.
6. Primary debulking surgery denied and maximum surgical effort of cytoreduction with the goal of no residual disease planned at interval debulking surgery. Sugarbaker index before inclusion must be less than 30
7. Eligible for carboplatin and paclitaxel chemotherapy in accordance with local standards of care following cy-toreductive surgery.
8. Interval complete surgery anticipated in a center with excellence.
9. ECOG performance status (PS) ≤ 2.
10. Life expectancy of at least 6 months,
11. Interval between diagnosis and enrolment (informed consent) ≤ 8 weeks,
12. Be willing to provide blood, and tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 8 weeks (56 days) prior to initiation of treatment on Day 1.
13. Demonstrate adequate organ function as defined in the table below, all screening labs should be performed within 7 days before randomization.
14. Adequate hematological laboratory value: Absolute neutrophil count (ANC): ≥1,500/mm3

    * Platelets : ≥100,000/mm3
    * Hemoglobin : ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
15. Adequate renal laboratory value:

    • Serum creatinine and Measured or calculated creatinine clearance a (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (Creatinine clearance is calculated according to Cockcroft formula or to MDRD formula for patients older than 65 years-old. Glo-merular filtration rate or creatinine clearance according to MDRD formula is: GFR = 186 x (creatinine (μmol/l) x 0,0113)-1,154 x age- 0,203 x 0.742.)
16. Adequate hepatic laboratory value:

    * Serum total bilirubin: ≤ 1.5 X ULN OR
    * Direct bilirubin: ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
    * LDH, CRP
    * AST (SGOT) and ALT (SGPT): ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
17. Adequate coagulation laboratory value:

    * International Normalized Ratio (INR) or Prothrombin Time (PT) : ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    * Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
18. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
19. Female subjects of childbearing potential should be willing to use 1 or 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 4 months after the last dose of study medication and 6 months after the last dose of bevacizumab, or paclitaxel, or carboplatin. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. (see below NB: contraception requirement)
20. Patient should be beneficiary of healthcare coverage under the social security system.

Exclusion Criteria:

1. Histological diagnosis of malignant tumor of non-epithelial origin (e.g. germ cell tumor, sex cord-stromal tumor) of the ovary, the fallopian tube or peritoneum or borderline tumor of the ovary (tumor of low malignant potential).
2. Patients with extra abdominal metastasis (FIGO 2014 Stage IV) not completely resectable, as e.g. multiple parenchymal lung metastases (preferably histologically proven), non resectable lymph node metastases, brain me-tastases.
3. Prior systemic therapy for ovarian cancer (e.g. chemotherapy, monoclonal antibody therapy, oral targeted therapy, hormonal therapy),
4. Prior radiotherapy to the abdomen or prior radiotherapy to an extra-abdominal target volume that would bear the risk of increased toxicity of chemotherapy,
5. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric or infectious disease, active ulcers (gastrointestinal tract, skin) or a laboratory abnormality that may Increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study,
6. Any contraindications for therapy with paclitaxel or carboplatin, e.g. a history of severe hypersensitivity reactions to paclitaxel or platinum-containing compounds and their excipients, or other drugs formulated with Pol-yoxyl 35Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
7. Diagnosis of immunodeficiency or receiving prolonged period of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
8. Known history of active Bacillus Tuberculosis (TB)
9. Hypersensitivity to pembrolizumab or any of its excipients.
10. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or no recovery (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
11. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
12. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. History of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Active Hepatitis B (e.g., HbsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Vaccination with a live vaccine within 30 days of planned start of study therapy.

    Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
18. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
19. Active infection requiring systemic therapy.
20. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule,
22. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Active alcohol or drug abuse,
24. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 4 months after the last dose of trial treatment, and six months after the last dose of bevacizumab, or paclitaxel, or carboplatin.
25. Patient unable to give their consent by their own (guardianship and curatorship)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Primary objective | Average of 4 months after the randomization of the last patient.
  Efficacy: Complete Resection Rate (CC0) after interval debulking surgery

SECONDARY OUTCOMES:
Secondary objective | Average of 4 months after the randomization of the last patient.
  Efficacy : CCI score evaluated by centers and by central review
Secondary objective | Average of 4 months after the randomization of the last patient.
  Efficacy : PCI score evaluated by centers and by central review
Secondary objective | Average of 4 months after the randomization of the last patient.
  Efficacy : Rate of Pathologic Complete Response (pCR) after surgery
Secondary objective | Average of 3 months after the first neo-adjuvant cycle.
  Efficacy : Objective Response Rate (ORR)
Secondary objective | From the date of randomization until the end of treatment.
  Efficacy : Best Overall Response
Secondary objective | From the date of randomization to date event, assessed up to 5 years.
  Efficacy : Progression-Free Survival (PFS)
Secondary objective | From the date of randomization to date event, assessed up to 5 years.
  Efficacy : Biological Progression-Free Interval (PFIBIO)
Secondary objective | From the date of randomization to death, assessed up to 5 years.
  Efficacy : Overall survival (OS)
Secondary objective | 30 days after last treatment intake.
  Safety and Tolerability of pembrolizumab in combination with chemotherapy : Incidence of Treatment-Emergent Adverse Events
Secondary objective | 30 days after the interval debulking surgery.
  Post-operative mortality
Secondary objective | 30 days after the interval debulking surgery.
  Post-operative morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle RAY-COQUARD, MD, PhD, Principal Investigator — isabelle.ray-coquard@lyon.unicancer.fr
Locations (22):
- France (22):
  - Hôpital Henri Duffaut, Avignon
  - CHRU Jean Minjoz, Besançon
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Groupe Hospitalier Diaconesses-Croix Saint Simon, Paris
  - Institut Mutualiste Montsouris-Jourdan, Paris
  - Centre CARIO-HPCA, Plérin
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - ICO Centre René Gauducheau, Saint-Herblain
  - CHU Saint-Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collet L, Ardin M, Venet D, Berthet J, Ghamry-Barrin S, Treilleux I, Noel JC, Leheurteur M, Meunier J, Bengrine Lefevre L, Martinez M, Priou F, Selle F, Just PA, Bataillon G, Rothe F, Sotiriou C, Caux C, Dubois B, Ray-Coquard I, Le Saux O. Unraveling the Tumor Microenvironment and PD-L1 Expression across Tissue Types in High-Grade Serous Ovarian Cancer in the NeoPembrOV/GINECO Phase II Randomized Trial. Clin Cancer Res. 2025 Aug 1;31(15):3317-3331. doi: 10.1158/1078-0432.CCR-24-2712. PMID 40378056
- See also: Acces to detailled results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-004163-39/results